CLINICAL TRIAL: NCT06237933
Title: Randomized Control Trial of a Social-networking-site(SNS) Based Weight Loss Behavior Intervention- the Effect of Social Network and Multi-level Factors on Weight Loss
Brief Title: A Social-networking-site(SNS) Based Weight Loss Behavior Intervention- the Effect of Social Network and Multi-level Factors on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201612183RINB
Record Dates: First submitted 2024-01-03; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced intervention (Experimental): Enhanced intervention features of using social-networking-site site and personalized feedback, plus standard intervention
  Interventions: Behavioral: Enhanced intervention via social networking site (SNS)
- Control (Active Comparator): Standard intervention with regular in-person consultation
  Interventions: Behavioral: Standard intervention

INTERVENTIONS:
Behavioral: Enhanced intervention via social networking site (SNS) — We plan to organize a private Facebook group serve as platform to provide the intervention content. To ensure confidentiality, this Facebook group is completely private and the group member is invited only by study staff. The participants of intervention group received information about the private Facebook group and privacy settings and were instructed to join the Facebook group. The intervention comprises three parts. Doctor patient interaction: The interventionist (physicians and dietitians) act as health coach will provide evidence-based topics related to weight loss on Facebook discussion board every two weeks
  Arms: Enhanced intervention
Behavioral: Standard intervention — In the session, the participants are instructed by an interventionist to have a reduced calorie diet and regular physical activity. Calorie intake was prescribed based on baseline weight at 1200 kcal/d for individuals who weighed less than 90 kg, 1500 kcal/d for those who weighed 90 to less than 115 kg, and 1800 kcal/d for those who weighed 115kg or more. The interventionist will give each participants dietary recommendation and sample meal plans are provided to facilitate adoption. The interventionist will prescribe non-supervised moderate-to-vigorous physical activity to participants. Participants should start moderate-to-vigorous physical activity at 100 minutes per week and increased at 4-week intervals until a prescription of 300 minutes per week was achieved
  Arms: Control

SUMMARY:
In this project, investigators plan to conduct a randomized control trial of a weight loss intervention that is remotely delivered via SNS among the obese adult patients (20-64 years old, BMI ≥ 27 kg/m2) recruited from weight control clinic in a tertiary medical center in Taipei. Investigators will survey the participants' baseline characteristics at different dimensions including personal, behavioral, physiological, socio-environmental factors. Participants will be randomly assigned to a 16-week weight loss program of either enhanced intervention via Facebook group or standard intervention. After the intervention, the participants will be followed until 2 years after enrollment. Investigators will measure participants' change in weight as well as change in attitude, behavior, and physiological along the follow-up periods. Investigators proposed specific study aims as following: (1) Demonstrate the characteristics of the obese patient who visiting weight-control clinics at behavioral level, physiological level, and social level. (2) Implement an enhanced weight loss intervention by using SNS with personalized feedback (3) Investigate the social influence and the interaction between participants in the social networking site (4) Test the hypothesis that, compared with a standard behavioral weight loss intervention, the enhanced intervention would result in greater weight loss and physical benefit (5) Test the hypothesis that, the enhanced intervention would result in improvement on heath attitude, literacy, or behavior and minimize the attrition of weight loss program (6) Explore the trajectory of individual characteristics throughout the treatment course (7) Explore the predictor or correlate of successful weight loss, maintenance and attrition (8) Investigate the interrelationship between different behavioral, physiological, and environmental factors and their composite effect on weight loss (9) Refine the intervention and develop a further effective and individualized behavior intervention for weight loss

DETAILED DESCRIPTION:
Obesity with its increasing prevalence has become a global health problem. Even modest weight loss induced by lifestyle intervention can produce clinically meaningful health benefits, however, most participants in the weight loss program fail in the longer term because of poor adherence and easy weight regain. An effective behavior therapy for weight loss is believed to have two core elements: (1) a convenient program focusing on individual response and variability, and (2) a better understanding of the predictors and correlates of weight loss outcome. Nowadays, the internet-based program featured with dynamic materials and personalized feedback has been utilized as a novel tool for weight loss. Besides, social networking site (SNS), such as Facebook, is a web-based platform for interaction. Increasing evidence demonstrated interventions through SNSs had substantial potentials on social influence and health behavior change. Research about the effectiveness of weight loss intervention via SNSs has gained much concern in recent years. Predictions of weight loss outcome based on personal characteristics are under investigation for several decades. Identifying predictors or correlates to weight loss outcome can help optimize the efficacy of the program through a better matching of intervention. Because weight loss is a is a dynamic and complex process encompassing interaction of behavioral, physiological and socio-environmental factors, a multi-factorial approach is required for research design. n this 3-year study project, investigators plan to conduct a pilot randomized control trial of a 2-year weight loss intervention that is remotely delivered via social networking site among the obese adult participants (20-64 years old, BMI ≥ 27 kg/m2) recruited from weight control clinic in medical center in Taipei, Taiwan. Investigators will survey the participants' baseline characteristics at different dimensions including personal, behavioral, physiological, social and environmental factors. Participants will be randomly assigned to a 16-week weight loss program of either enhanced intervention via Facebook or standard intervention. After the intervention, the participants will be followed for another 1 year and 8 months. The change in weight will be measured at 6 months, 12 months and 24 months after enrollment. Participants' change in attitude, behavior, and physiological condition will also be measured along the follow-up so that investigators can demonstrate the trajectory and interaction of different variables along the weight loss process. With this 3-year project, investigators not only assess the efficacy of this pilot weight loss program in Taiwan, but investigators also explore the possible predictors and correlates of successful weight loss.

ELIGIBILITY:
Inclusion criteria:

* Aged 20-64 years
* Body mass index (BMI) ≥27 kg/m2
* Used Facebook or were willing to begin, owned a personal computer or owned a smartphone, and are healthy enough and willing to attend this program with measurement visits in 2 years.

Exclusion criteria:

* Pregnancy
* Previous diagnosis of diabetes mellitus
* History of psychosis, severe anxiety, major depression, panic, or Clinically diagnosed eating disorder
* History of surgical treatment for obesity
* Alcoholism or drug abuse.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
weight change | 4weeks, 8weeks, 13weeks, 26weeks, 52weeks, 78weeks, 104weeks
  Weight in kilogram is assessed to the nearest 0.1 kg with the participant clothed in lightweight clothing. Weight change is calculated as weight after intervention minus weight at baseline. Weight change is calculated for each participant.

SECONDARY OUTCOMES:
Participants' eating behavior | 26weeks, 52weeks, 78weeks, 104weeks
  The questionnaire, three factor eating questionnaire-R18(TFEQ-R18), for assessment of participants' eating behavior. (The minimum score of TFEQ-R18 for eating behavior I(cognitive restraint of eating)-II(disinhibition)-III(hunger) is therefore 0-0-0, and maximum possible score is 20-16-15. Higher score means higher tendency of each eating behavior).
Participants' psychological distress | 26weeks, 52weeks, 78weeks, 104weeks
  The questionnaire, Brief Symptom Rating Scale-5(BSRS-5) for assessment of participants' psychological distress. (The minimum score of BSRS-5 is 0 and maximum possible score is 20. Higher score means worse outcome, higher psychological distress.)
Participants' quality of life | 26weeks, 52weeks, 78weeks, 104weeks
  The questionnaire, Clinical Impairment Assessment Questionnaire(CIA 3.0) for assessment of participants' quality of life. (The minimum score of CIA 3.0 is 0 and maximum possible score is 48. Higher score means worse outcome, poor quality of life.)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No